CLINICAL TRIAL: NCT01009671
Title: Randomised, Comparative, Double-blind, Parallel-group Study to Evaluate the Digestive Tolerability of ART44 Versus ART®50 in Patients With Osteoarthritis of the Knee
Brief Title: Study to Evaluate the Digestive Tolerability of ART44 Versus ART®50 in Patients With Osteoarthritis of the Knee
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Laboratoires NEGMA (Industry)
Responsible Party: Patrick DARSES, Laboratoires NEGMA
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HEC/ARTGT/081000N; 2009-009990-84
Record Dates: First submitted 2009-11-06; First posted 2009-11-09 (Estimated); Last update posted 2009-11-09 (Estimated); Status verified 2009-11

CONDITIONS: Knee Osteoarthritis
Keywords: knee osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- ART 44 (Experimental): Evaluation of safety and efficacy at D-8, D0, W2, W4 and W12
  Interventions: Drug: ART 44
- ART 50 (Active Comparator): Evaluation of safety and efficacy at D-8, D0, W2, W4 and W12
  Interventions: Drug: ART 50

INTERVENTIONS:
Drug: ART 44
  Arms: ART 44
Drug: ART 50
  Arms: ART 50

SUMMARY:
The primary objective of this study, comparing ART 44 to ART 50, will be the evaluation of digestive tolerability (and in particular of diarrhoea).

ELIGIBILITY:
Inclusion Criteria:

* Female or Male, aged 40 to 80 years, outpatient;
* Presenting with internal femorotibial osteoarthritis:

  * Symptomatic for more than 6 months;
  * Meeting ACR clinical and radiological criteria;
  * Overall mean VAS score of knee pain in last 24 hours > 40 mm (with no NSAIDs for over 72 hours and no analgesics for over 24 hours);
  * Pain present for at least one day out of 2 in the month preceding enrolment;
  * Radiological stage II to III (Kellgren and Lawrence) (image less than 12 months old).

Exclusion Criteria:

* Associated predominant symptomatic femoropatellar osteoarthritis;
* Chondromatosis or villonodular synovitis of the knee;
* Paget's Disease.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2009-11; Primary Completion 2010-08 (Estimated); Study Completion 2010-10 (Estimated)

PRIMARY OUTCOMES:
To demonstrate the better digestive tolerability of ART44 versus ART 50 over a 1-month period, based on a clinically predetermined difference | Day 8, Day 0, Week 2, Week 4 and Week 12

SECONDARY OUTCOMES:
To compare the overall safety and efficacy of the two products | Day 8, Day 0, Week 2, Week 4 and Week 12